CLINICAL TRIAL: NCT01138917
Title: A Multicenter Comparative Study of the ReCell Device and Autologous Split-thickness Meshed Skin Graft in the Treatment of Acute Burn Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avita Medical (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency); Royal Perth Hospital (Other); MedDRA Assistance Inc (Unknown); BioStat International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTP001-5
Record Dates: First submitted 2010-06-03; First posted 2010-06-08 (Estimated); Results first posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Burns
Keywords: Second Degree Burn Injuries
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- all participants (Experimental): All participants will receive both ReCell and split-thickness skin graft
  Interventions: Device: ReCell and Split-thickness skin graft

INTERVENTIONS:
Device: ReCell and Split-thickness skin graft — The surgeon will be required to select two similar non-contiguous injury areas with both areas being at least 100cm2 and second degree depth/severity. One area will be treated using ReCell and the second using Split-thickness Skin Graft.

SUMMARY:
This is a randomized, within-patient controlled study to compare the clinical performance of the ReCell Device with that of Split-thickness Meshed Skin Grafts for the treatment of second degree burns. The hypothesis to be supported are: 1) non-inferiority with the primary efficacy endpoint defined as recipient site wound closure at week 4 follow-up visit of the ReCell-treated area as compared to that of the STMSG-treated area, and 2)superiority in the healing of the ReCell donor site as compared to the STMSG donor site at week 1.

ELIGIBILITY:
Inclusion Criteria:

* The subject requires primary skin grafting as a result of an acute thermal burn injury
* The area of the burn injury is at least 200cm2 (1% TBSA in adults) if a contiguous wound, or at least 100cm2 for each of 2 noon-contiguous wounds
* The area of total burn injury is 1-20% TBSA
* The burn injured area can be divided into two treatment areas ( control and treatment) with 100-320cm2 area for each treatment type
* The study treatment area is a second degree burn injury
* The subject is between 18-65 years of age
* The subject is willing to complete all follow-up evaluations required by the study protocol
* The subject is to abstain from any other treatment of the wound(s) for the duration of the study unless medically necessary
* The subject agrees to abstain from enrollment in any other clinical trial for the duration of the study
* The subject and/or guardian are able to read and understand instructions and give informed, voluntary, written consent
* The subject is able and willing to follow the protocol requirements

Exclusion Criteria:

* The subject's burn injuries were caused by chemicals, electricity, and/or radioactive substances
* The total subject burn injury is less than 1% or more than 20% TBSA
* The subject has a microbiologically proven pre-existing local or systemic bacterial infection
* The subject has been receiving a systemic antibiotic for more than 48 hours prior to grafting
* The subject is known to have a pre-existing condition that may interfere with wound healing ( e.g. malignancy, diabetes, or autoimmune disease)
* The subject is unable to follow the protocol
* The subject is taking medication known to have an effect on wound healing or skin pigmentation ( e.g. systemic corticosteroids, retinoids, etc)
* The subject has other concurrent conditions that in the opinion of the investigator may compromise patient safety or study objectives
* The subject has a known hypersensitivity to Trypsin or Compound sodium Lactate for Irrigation (Hartmann's) solution

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2010-05-21 (Actual); Primary Completion 2014-08-29 (Actual); Study Completion 2015-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James H Holmes, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (12):
- United States (12):
  - Arizona Burn Center at Maricopa Integrated Health Systems, Phoenix, Arizona
  - University of California Davis Regional Burn Center, Sacramento, California
  - The Burn Center at Washington Hospital Center, Washington D.C., District of Columbia
  - Shands Burn Center at University of Florida, Gainesville, Florida
  - Tampa General Hospital, Tampa, Florida
  - Indiana University - Richard M. Fairbanks Burn Center at Wishard Memorial Hospital, Indianapolis, Indiana
  - NC Jaycee Burn Center at University of NC at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Tennessee Medical Center, Memphis, Tennessee
  - USAISR, Fort Sam Houston, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Virginia Commonwealth University Health System- Evans Haynes Burn Center, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: All Participants (Within Patient Control): Every subject received both interventions (RECELL and Control (2:1 meshed split-thickness autograft)). Two distinct but similar areas of burn injury at least 100 cm2 and second degree depth will be treated according to random assignment (Area A and Area B). One burn injury area receives RECELL (Investigational Treatment) and the other area Control (2:1 meshed autograft).
Period: Overall Study
Arm/Group | Experimental: All Participants (Within Patient Control)
Started | 101
Completed | 77
Not Completed | 24

BASELINE CHARACTERISTICS:
Groups:
- Experimental: All Participants (Within Patient Control): Every subject received both interventions (RECELL and 2:1 meshed split-thickness autograft). Two distinct but similar areas of burn injury at least 100 cm2 and second degree depth will be treated according to random assignment (Area A and Area B). One burn injury area receives RECELL (Investigational Treatment) and the other area 2:1 meshed autograft (Control).
Arm/Group | Experimental: All Participants (Within Patient Control)
Number analyzed (Participants) | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 101
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (13.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 85
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 59
  Race: Hispanic | 19
  Race: Asian | 1
  Race: American Indian | 0
  Race: Black | 20
  Race: Other | 2
Region of Enrollment [Number; unit: participants]
  United States | 101

OUTCOME MEASURES:

1. Primary Outcome: Incidence of RECELL-treated Area Closure Compared to Control at 4 Weeks (Non-inferiority)
Description: Recipient site wound closure for both ReCell and STMSG will be defined as the presence of >=95% epithelialization with contiguous layer of viable epithelium without the need for secondary surgical intervention. Factors considered during the assessment included color, presence of granulation tissue, and whether or not the entire wound is covered with a contiguous layer of viable epithelium. Using this definition, some small degree of punctate blistering was acceptable as long as the wound was >=95% epithelialized.
Time Frame: 4 weeks
Population: Analysis to evaluate non-inferiority of recipient site wound closure was performed on the ITT, PP, and MPP populations.
Measure: Count of Participants; unit: Participants
Groups:
- RECELL: Cell suspension prepared using the RECELL device applied to "RECELL Recipient Site"
- Control: 2:1 meshed autograft applied to "Control Recipient Site"
Arm/Group | RECELL | Control
Number analyzed (Participants) | 101 | 101
Participants
  Per Protocol Population (PP): number analyzed (Participants) | 87 | 87
  Per Protocol Population (PP) | 82 | 87
  Modified Per Protocol Population (MPP): number analyzed (Participants) | 83 | 83
  Modified Per Protocol Population (MPP) | 82 | 83
  Intent to Treat (ITT) | 84 | 97

2. Primary Outcome: Incidence of RECELL Donor Site Healing Compared to Control at 1 Week (Superiority)
Description: Donor site healing will be considered as complete (100%) wound closure if the following criteria were met: an ability to separate the dressing from the wound bed with visible presence over the entirety of the wound of dry, opalescent-pink external surface representing the newly formed outer cornfield layer of the epidermis.
Time Frame: 1 week
Population: Analysis was performed on ITT, PP, and MPP populations. Note: The number of participants with evaluable donor sites differs than number of participants with evaluable recipient sites.
Measure: Count of Participants; unit: Participants
Groups:
- RECELL: RECELL donor site
- Control: Control donor site
Arm/Group | RECELL | Control
Number analyzed (Participants) | 100 | 100
Participants
  Intent to Treat (ITT) | 22 | 10
  Per Protocol (PP): number analyzed (Participants) | 88 | 88
  Per Protocol (PP) | 19 | 10
  Modified Per Protocol (MPP): number analyzed (Participants) | 82 | 82
  Modified Per Protocol (MPP) | 18 | 10

3. Secondary Outcome: Percent of Epithelialization at Each Visit Through Week 16
Description: The percent epithelialization of the RECELL and Control treated sites will be assessed using standardized planimetry/tracing procedures. The tracings were uploaded to a Central Reading Facility for calculation of percent epithelialization using a computerized measurement technique.
Time Frame: Each visit through Week 16
Population: Percent Epithelialization presented for Per Protocol Population (PP) based on subjects presented for healing evaluation per visit
Measure: Mean (Standard Deviation); unit: percentage of epithelialization
Arm/Group | RECELL | Control
Number analyzed (Participants) | 87 | 87
percentage of epithelialization
  % Epithelialization - Week 1: number analyzed (Participants) | 83 | 84
  % Epithelialization - Week 1 | 66.1 (40.94) | 74.0 (41.25)
  % Epithelialization - Week 2 | 92.1 (20.38) | 99.8 (1.16)
  % Epithelialization - Week 3: number analyzed (Participants) | 84 | 85
  % Epithelialization - Week 3 | 95.8 (14.90) | 99.9 (0.58)
  % Epithelialization - Week 4 | 97.7 (11.98) | 100.0 (0.07)
  % Epithelialization - Week 8: number analyzed (Participants) | 86 | 86
  % Epithelialization - Week 8 | 99.8 (1.42) | 100.0 (0.00)
  % Epithelialization - Week 16 | 100.0 (0.00) | 100.0 (0.00)

4. Secondary Outcome: Wound Closure at Week 2 (Based on Investigators Assessment)
Description: The proportion of recipient sites achieving wound closure at Week 2 was evaluated using the Investigators assessment of wound healing.
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Groups:
- Recipient Site Wound Healing at Week 2: Investigator Assessment of Recipient Site Wound Healing Per-Protocol Population
Arm/Group | Recipient Site Wound Healing at Week 2
Number analyzed (Participants) | 87
Participants
  RECELL and Control Healed | 70
  RECELL Healed and Control Not Healed | 1
  RECELL Not Healed and Control Healed | 16
  RECELL and Control Not Healed | 0

5. Secondary Outcome: Mean Pain and Appearance Scores at RECELL and Control Recipient Sites (Subject Assessment)
Description: Subject assessment of pain at the RECELL and Control recipient sites was performed at all study follow-up visits up to Week 16.
  Subjects also assessed the satisfaction with the appearance of the treatment sites at the Week 16, 24, and 52 study follow-up visits. The subject assessments were performed using VAS (visual analogue scale) style questionnaires.
  Pain VAS 0-100 where 0=non-existent pain and 100=severe pain. Appearance VAS 0-100 where 0=terrible and 100=exceptional
Time Frame: Pain (Weeks 1-16) and Appearance (Weeks 16-52)
Population: Per-Protocol Population
Measure: Mean (Standard Deviation); unit: Scores on a Scale (0-100)
Arm/Group | RECELL | Control
Number analyzed (Participants) | 87 | 87
Scores on a Scale (0-100)
  Mean Pain Scores at Week 1: number analyzed (Participants) | 80 | 80
  Mean Pain Scores at Week 1 | 24.1 (23.31) | 26.5 (24.58)
  Mean Pain Scores at Week 2: number analyzed (Participants) | 85 | 85
  Mean Pain Scores at Week 2 | 12.4 (19.42) | 12.4 (19.10)
  Mean Pain Scores at Week 3: number analyzed (Participants) | 85 | 85
  Mean Pain Scores at Week 3 | 9.6 (14.39) | 7.9 (14.60)
  Mean Pain Scores at Week 4 | 6.9 (12.64) | 6.7 (12.25)
  Mean Pain Scores at Week 8: number analyzed (Participants) | 86 | 86
  Mean Pain Scores at Week 8 | 7.6 (16.94) | 8.8 (18.46)
  Mean Pain Scores at Week 16: number analyzed (Participants) | 81 | 81
  Mean Pain Scores at Week 16 | 3.3 (8.15) | 4.3 (10.56)
  Mean Visual Appearance Week 16: number analyzed (Participants) | 83 | 83
  Mean Visual Appearance Week 16 | 77.7 (23.96) | 75.6 (24.18)
  Mean Visual Appearance Week 24: number analyzed (Participants) | 72 | 72
  Mean Visual Appearance Week 24 | 82.6 (22.82) | 79.4 (22.78)
  Mean Visual Appearance Week 52: number analyzed (Participants) | 70 | 70
  Mean Visual Appearance Week 52 | 83.1 (22.07) | 80.1 (19.73)

6. Secondary Outcome: Mean Pain and Appearance Scores at Donor Sites (Subject Assessment)
Description: Subject assessment of pain at the RECELL and Control donor sites was performed at all study follow-up visits up to Week 16.
  Subjects also assessed the satisfaction with the appearance of the donor sites at the Week 16, 24, and 52 study follow-up visits. The subject assessments were performed using VAS (visual analogue scale) style questionnaires.
  Pain VAS 0-100 where 0=non-existent pain and 100=severe pain. Appearance VAS 0-100 where 0=terrible and 100=exceptional.
Time Frame: Pain (Weeks 1-16) and Appearance (Weeks 16-52)
Population: Per-Protocol Population
Measure: Mean (Standard Deviation); unit: Scores on a Scale (0-100)
Arm/Group | RECELL | Control
Number analyzed (Participants) | 87 | 87
Scores on a Scale (0-100)
  Mean Pain Scores at Week 1: number analyzed (Participants) | 80 | 80
  Mean Pain Scores at Week 1 | 21.9 (26.35) | 43.5 (29.43)
  Mean Pain Scores at Week 2: number analyzed (Participants) | 85 | 85
  Mean Pain Scores at Week 2 | 5.1 (11.25) | 19.3 (24.42)
  Mean Pain Scores at Week 3: number analyzed (Participants) | 85 | 85
  Mean Pain Scores at Week 3 | 1.9 (3.87) | 9.4 (19.14)
  Mean Pain Scores at Week 4 | 1.9 (5.84) | 5.2 (12.07)
  Mean Pain Scores at Week 8: number analyzed (Participants) | 86 | 86
  Mean Pain Scores at Week 8 | 1.4 (2.78) | 3.7 (9.97)
  Mean Pain Scores at Week 16: number analyzed (Participants) | 81 | 81
  Mean Pain Scores at Week 16 | 0.9 (1.61) | 1.5 (2.84)
  Mean Visual Appearance Week 16: number analyzed (Participants) | 83 | 83
  Mean Visual Appearance Week 16 | 89.8 (16.87) | 75.1 (26.36)
  Mean Visual Appearance Week 24: number analyzed (Participants) | 72 | 72
  Mean Visual Appearance Week 24 | 93.4 (9.96) | 81.1 (21.55)
  Mean Visual Appearance Week 52: number analyzed (Participants) | 70 | 70
  Mean Visual Appearance Week 52 | 91.2 (14.84) | 83.3 (18.62)

ADVERSE EVENTS:
Time Frame: All adverse events occurring during the course of the clinical study were reported. Adverse event reporting was limited to wound findings, i.e. scarring, contraction, etc. of the study wound areas at Week 16 through to Week 52.
Description: The number of specific adverse events that occurred per wound area is included in the Adverse Event Term Additional Description.
Groups:
- Experimental: All Participants (Within Patient Control): All subjects received cell suspension prepared using the RECELL device applied to "RECELL Recipient Site" and 2:1 meshed conventional autografting applied to "Control Recipient Site"
Arm/Group | Experimental: All Participants (Within Patient Control)
Serious Adverse Events (participants affected / at risk) | 10/101
Other Adverse Events (participants affected / at risk) | 34/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: All Participants (Within Patient Control) (N=101)
Nausea, Vomiting, Diarrhea (Gastrointestinal disorders) | 1 (1)
Blood clot detected in left leg (Vascular disorders) | 1 (1)
Scar contracture release (Injury, poisoning and procedural complications) | 1 (1) — Other wound
>10% graft loss (Injury, poisoning and procedural complications) | 1 (1) — RECELL Recipient Site
Burn wound excision/grafting (Injury, poisoning and procedural complications) | 1 (1) — Other wound
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
New burn injury (Injury, poisoning and procedural complications) | 1 (1) — RECELL Recipient Site
New burn injury (Injury, poisoning and procedural complications) | 1 (1) — Control Recipient Site
Suspected wound infection (Infections and infestations) | 1 (1) — RECELL Recipient Site
Graft failure conversion to full thickness wound (Injury, poisoning and procedural complications) | 1 (1) — RECELL Recipient Site
Coumadin toxicity (Injury, poisoning and procedural complications) | 1 (1)
Worsening anemia post-operatively (Blood and lymphatic system disorders) | 1 (1)
Intraoperative tachycardia resolved with fluids and beta-blockade (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: All Participants (Within Patient Control) (N=101)
Hypertrophic Scar (Skin and subcutaneous tissue disorders) | 15 (26) — RECELL Recipient Site (n=10) Control Recipient Site (n=6) Other (n=11)
Rash (Skin and subcutaneous tissue disorders) | 5 (6) — RECELL Recipient Site (n=3) Control Recipient Site ((n=1) Other (n=2)
Hypergranulated Tissue/Hypergranulation (Skin and subcutaneous tissue disorders) | 7 (10) — RECELL Recipient Site (n=8) Control Recipient Site (n=1) Other (n=1)
Itching/Pruritus (Skin and subcutaneous tissue disorders) | 6 (14) — RECELL Recipient Site (n=5) Control Recipient site (n=5) Other (n=4)
Hypertrophy (General disorders) | 7 (13) — RECELL Recipient Site (n=5) Control Recipient Site (n=3) Other (n=5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No